CLINICAL TRIAL: NCT04470206
Title: Spinal Cord Stimulation for Neuropathic Pain Relief : Efficacy Study Using the Specific NPSI Questionnaire
Brief Title: Spinal Cord Stimulation for Neuropathic Pain Relief : Efficacy Study Using the Specific NPSI Questionnaire (NPSI)
Acronym: NPSI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_0080
Record Dates: First submitted 2020-07-08; First posted 2020-07-14 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Neuropathic Pain
Keywords: Neuropathic pain; NPSI; Spinal Cord Stimulation
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Several studies have shown the efficacy of spinal cord stimulation in reducing the intensity of neuropathic pain. This efficacy is defined as obtaining relief of at least 50% of the preoperative pain intensity assessed by the visual analog scale or the digital pain scale. No study has evaluated the efficacy of stimulation specifically on the different components of neuropathic pain, only an overall improvement in pain has been described.

A specific questionnaire for neuropathic pain has been extensively validated in neuropathic pain: the Neuropathic Pain Symptom Inventory (NPSI).

Thanks to the multidimensional structure of this questionnaire, investigators propose to evaluate separately and in a much more specific way the efficacy of spinal cord stimulation in the short and long term on the different components of neuropathic pain and to define responders subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* With neuropathic pain:

  * confirmed (DN4 score> 4/10)
  * going back to one year at least
  * refractory to well-conducted medical treatments
* Requiring spinal cord stimulation: the indication is validated by the multidisciplinary meeting (RCP Neuromodulation / Pain at Foch Hospital)
* Having given his non-opposition

Exclusion Criteria:

* Patient with sepsis
* Having no well-conducted prior medical treatment
* With uncontrolled psychiatric disorders (active psychosis, suicidal disorders, severe depression)
* with somatoform disorders
* addicted to alcohol or drugs or withdrawal syndrome
* Deprived of liberty or under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neuropathic pain following surgery or in the context of a complex regional pain syndrome and requiring spinal cord stimulation in the neurosurgery department of Foch Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10-19 (Actual); Primary Completion 2023-12-19 (Estimated); Study Completion 2023-12-19 (Estimated)

PRIMARY OUTCOMES:
Efficacy of spinal cord stimulation on the various symptoms of neuropathic pain using the Neuropathic Pain Symptom Inventory (NPSI), change is being assessed. | Day 0; Day 7 after surgery; 3 months, 6 months and 12 months after surgery
  Neuropathic pain score obtained by the NPSI questionnaire

SECONDARY OUTCOMES:
Efficacy of spinal cord stimulation on the psychological level (anxiety and depression) | Day 0 and 12 months after surgery
  Anxiety and depression score assessed by Hospital Anxiety and Depression (HAD) questionnaire
Efficacy of spinal cord stimulation on quality of life. | Day 0 and 12 months after surgery
  Quality of life score assessed by EQ-5D questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Naoufel Ouerchefani, MD, Principal Investigator — Foch Hospital
Locations (1):
- Hôpital Foch, Suresnes, Île-de-France Region, France